CLINICAL TRIAL: NCT07095634
Title: Protocollo Sulla Valutazione Del RischiO cardioVAscolare Nel Crohn e ColIte Ulcerosa (PROVACI). Estimation of Cardiovascular Risk in Crohn's Disease and Ulcerative Colitis
Brief Title: Estimation of Cardiovascular Risk in Patients With Crohn's Disease and Ulcerative Colitis (PROVACI)
Acronym: PROVACI
Status: Enrolling by invitation | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Vito Annese, Associate Professor University Vita-Salute San Raffaele, Milan; Head of Gastroenterology IRCCS San Donato Policlinic, IRCCS Policlinico S. Donato
Other Study IDs: CET 510-2024
Record Dates: First submitted 2025-07-23; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Ulcerative Colitis; Myocardial Infarction; Stroke; Ischemic Heart Disease; Atrial Fibrillation (AF); Thromboembolism; Crohn Disease; Transient Ischemic Attack (TIA); Heart Failure
Keywords: Cardiovascular risk in IBD
MeSH Terms: conditions — Colitis, Ulcerative; Myocardial Infarction; Stroke; Myocardial Ischemia; Atrial Fibrillation; Thromboembolism; Crohn Disease; Ischemic Attack, Transient; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood sample, biopsies and stool
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBD Patients (either with Crohn's disease or ulcerative colitis): Baseline evaluation of CV risk score + comprehensive clinical characteristics
- Control subjects without IBD: Age-and gender-matched cohort under cardiologic follow-up

SUMMARY:
Inflammatory bowel diseases (IBD) are progressively increasing their prevalence worldwide. Up to half of patients may also have extraintestinal manifestation and cardiovascular diseases (CVDs) is one of the most relevant, being the second cause of death in these patients. The classical cardiovascular (CV) risk scores do not adquately capture the CV risk in IBD.

We are planning a prospective observational study to evaluate patients with IBD and a gender/age-matched cohort with the aims to investigate in 2-years follow-up

* Occurrence of major cardiovascular events (MACEs) in both cohorts;
* Predictive factors of risk for MACEs in IBD compared to controls;
* Multi-omics evaluations with the support of artificial intelligence of biomarkers associated with occurrence of MACEs in IBD

ELIGIBILITY:
Inclusion Criteria:

Patients with confrimed diagnosis of Crohn's disease and Ulcerative colitis-

Exclusion Criteria:

No willing to sign the informe content and have 2 years of follow-up

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: IBD patients willing to remain in follow-up for 2 years
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Major cardiovascular events | 2 years
  Myocardial infarction, stroke, transient ischemic attack, heart failure, atrial fibrillation, acute arterial embolysm, ischemic angina

SECONDARY OUTCOMES:
Multi-omics evaluations of biomarkers in IBD patients with occurrence of MACEs | 2 years follow-up
  Genomics - genetics score of investigated variants Transcritptomics - gene expression different in IBD patients with and without MACEs Microbiome - difference among IBD patients with and without MACEs Combined analysis of multi-omics data set and clinical characteristics with artificial intelligence

CONTACTS AND LOCATIONS:
Overall Officials: Vito Annese, Prof, Principal Investigator — IRCCS Policlinico San Donato, Universita' Vita-Salute San Raffeele, Milano, Italy
Locations (1):
- IRCCS San Donato POliclinic, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Characteristics of Study and control cohorts
Supporting Information: Study Protocol, ICF, CSR
Time Frame: At the end of Follow-up (End of 2028). It will be available for 5 years
Access Criteria: Any researcher, provided that will have an approved scientific plan to gather clinical info of the study (IBD) and control cohorts
URL: https://www.google.com/url?sa=t&source=web&rct=j&opi=89978449&url=https://www.grupposandonato.it/strutture/policlinico-san-donato/contatti&ved=2ahUKEwi5sIL2_9KOAxXCiP0HHfV1JHAQFnoECBwQAQ&usg=AOvVaw2nNbGXySjQHZH9GVwkP1sN